CLINICAL TRIAL: NCT03467737
Title: Assessing Malian and U.S. Children for Starch Digestion and Amylase Sufficiency and Identifying Better Energy Providing Foods for Growth and Recovery
Brief Title: Assessment of Starch Digestibility and Amylase Sufficiency in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1209012695
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — octanoic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Normal sorghum porridge, algal starch (Experimental): Sorghum porridge with 13C-algal starch
  Interventions: Other: Normal sorghum porridge, algal starch
- Normal sorghum porridge, algal dextrins (Experimental): Sorghum porridge with 13C-algal starch limit dextrins
  Interventions: Other: Normal sorghum porridge, algal dextrins
- Normal sorghum porridge, labeled flour (Experimental): Sorghum porridge with 13C-labeled sorghum flour
  Interventions: Other: Normal sorghum porridge, labeled flour
- Modified sorghum porridge, labeled flour (Experimental): Modified sorghum porridge with 13C-labeled sorghum flour
  Interventions: Other: Modified sorghum porridge, labeled flour
- Thinned sorghum porridge, labeled flour (Experimental): Modified thinned sorghum porridge with 13C-labeled sorghum flour
  Interventions: Other: Thinned sorghum porridge, labeled flour
- Modified sorghum porridge, octanoic acid (Experimental): Modified sorghum porridge with 13C-labeled octanoic acid
  Interventions: Other: Modified sorghum porridge, octanoic acid

INTERVENTIONS:
Other: Normal sorghum porridge, algal starch — Normal sorghum porridge with 13C-labeled algal starch was fed, breath tested, as the first arm of an alpha-amylase sufficiency assessment in healthy and moderately malnourished children.
  Arms: Normal sorghum porridge, algal starch
Other: Normal sorghum porridge, algal dextrins — Normal sorghum porridge with 13C-labeled starch limit dextrins was fed, breath tested, as the second arm of an alpha-amylase sufficiency assessment in healthy and moderately malnourished children.
  Arms: Normal sorghum porridge, algal dextrins
Other: Normal sorghum porridge, labeled flour — Normal sorghum porridge with a portion of 13C-labeled sorghum flour was fed, breath tested, for starch digestibility assessment in healthy and moderately malnourished children.
  Arms: Normal sorghum porridge, labeled flour
Other: Modified sorghum porridge, labeled flour — Modified sorghum porridge with shear stirring to reduce viscosity with a portion of 13C-labeled sorghum flour was fed, breath tested, for starch digestibility assessment in healthy and moderately malnourished children.
  Arms: Modified sorghum porridge, labeled flour
Other: Thinned sorghum porridge, labeled flour — Thinned sorghum porridge treated with an alpha-amylase liquifying enzyme with a portion of 13C-labeled sorghum flour was fed, breath tested, for starch digestibility assessment in healthy and moderately malnourished children.
  Arms: Thinned sorghum porridge, labeled flour
Other: Modified sorghum porridge, octanoic acid — Modified sorghum porridge with shear stirring to reduce viscosity with addition of 13C-labeled octanoic acid was fed, breath tested, for gastric emptying assessment in healthy and moderately malnourished children.
  Arms: Modified sorghum porridge, octanoic acid

SUMMARY:
Research has demonstrated that there is a relationship between malnourishment and insufficient production of pancreatic enzymes, such as α-amylase which digests starch into glucose. Starchy foods that can be easily digested into glucose are critical to the development child for energy and proper growth. This study investigated the use of a noninvasive breath test for the assessment of amylase sufficiency, digestibility of normal and modified sorghum porridges and gastric emptying rate of a sorghum porridge in Malian and U.S. children.

DETAILED DESCRIPTION:
The purpose of this research is to test the hypotheses that: 1.) Moderately malnourished stunted children have low pancreatic α-amylase activity; and 2.) Modified starchy food preparations will have better (higher) digestibility than the commonly given foods for both moderately malnourished stunted and healthy non-stunted children. A noninvasive breath test was used to assess amylase insufficiency in moderately malnourished and stunted children in Mali, as well as in healthy children in Mali and the United States. Moderately malnourished and healthy children in Mali were fed sorghum porridges, which are commonly consumed in Mali. Porridges contained a 13C-labeled substrate (algal starch or octanoic acid) for assessment of amylase insufficiency and gastric emptying rate. In a follow-up study, healthy children in the United States were also assessed for amylase sufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Stunted weaned children in the age range 18 - 30 months with height-for-age Z-score (HAZ) below -2 (HAZ<-2)
* Healthy, weaned children 18-30 months of age for study 1
* Healthy, weaned children up to 5 years old

Exclusion Criteria:

* Acutely ill and wasted child with weight for height lower than -2 z-score
* No medical problems other than their malnutrition status
* No medications

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Alpha-amylase sufficiency in children | 3 hours after being fed test meal
  Breath test using 13C-tracer was used to assess alpha-amylase sufficiency in healthy and moderately malnourished children
Starch digestibility | 3 hours after being fed test meal
  Breath test using 13C-tracer in labeled sorghum flour was used to assess starch digestibility of three different prepared sorghum porridges of different thicknesses in healthy and moderately malnourished children
Gastric emptying | 3 hours after being fed test meal
  Breath test using 13C-tracer in octanoic acid was used to assess gastric emptying in healthy and moderately malnourished children

IPD SHARING:
Plan to Share IPD: No
Not shared